CLINICAL TRIAL: NCT04004000
Title: An Open-Label Pilot Study of Losmapimod to Evaluate the Safety, Tolerability, and Changes in Biomarker and Clinical Outcome Assessments in Subjects With Facioscapulohumeral Muscular Dystrophy 1 (FSHD1) With Extension
Brief Title: Evaluation of Safety, Tolerability, and Changes in Biomarker and Clinical Outcome Assessments of Losmapimod for FSHD1 With Extension
Acronym: FSHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIS-001-2019
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Facioscapulohumeral Muscular Dystrophy 1
Keywords: FSHD, FSHD1; Muscular Dystrophies; Facioscapulohumeral Muscular Disorders; Atrophic Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Intervention Model Description: This is a single-centre, open-label pilot study with open-label extension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): FSHD1 subjects with genetic confirmation will receive 15 mg of losmapimod twice daily given by mouth; for a total of 30 mg daily until 90 days after commercial drug is available post regulatory approval or study termination.
  Interventions: Drug: Losmapimod

INTERVENTIONS:
Drug: Losmapimod — The main study includes a treatment period of approximately one year. Subjects will receive 15 mg of losmapimod twice daily by mouth; for a total of 30 mg daily. The study drug should be taken with food and the date and time of each dose taken recorded in the subject diary.
  Only subjects who participated in and completed all procedures for the main study (Week 60) will be eligible to participate in the extension.
  For the extension, subjects will receive 15 mg of losmapimod by mouth twice daily for a total of 30 mg by mouth daily. Participation will continue until 90 days after commercial drug is available post regulatory approval or study termination.

SUMMARY:
This clinical trial is a study to evaluate the safety, tolerability, and changes in biomarker and clinical outcome assessments of Losmapimod for patients with Facioscapulohumeral Muscular Dystrophy 1 (FSHD1) with an open-label extension.

DETAILED DESCRIPTION:
This study is a single-centre, open-label pilot study that will investigate the safety, tolerability, pharmacokinetics (PK), and target engagement during long-term dosing with losmapimod tablets in adult subjects with FSHD1. Subjects will be evaluated during an 8- week pre-treatment period (Visits 1 through 3) to establish pre-treatment baseline assessments. Subjects will then be treated with losmapimod for approximately 1 year (Visits 4 through 9) and assessed at relatively regular intervals for change from pre-treatment assessments. All subjects will undergo two muscle biopsies; one at baseline, pre-treatment (Visit 4, Week 8 ± 1 week) and the second on-treatment muscle biopsy approximately 4 or 8 weeks later (Visit 5, Week 14 ± 2 weeks). Up to 8 subjects will have an on-treatment biopsy at 4 weeks and up to 8 subjects will have the on-treatment biopsy at 8 weeks.

Only subjects who participated in and competed all study procedures in the OLS Study treatment period (Week 60) will be eligible to participate in the open-label extension study.

The extension of this study will enable continued investigation of the safety and tolerability of long-term dosing with losmapimod tablets in adult subjects with FSHD1. During the extension study, subjects will receive 15 mg of losmapimod by mouth twice daily for a total of 30 mg by mouth daily. All subjects will attend clinic visits approximately every 24 weeks and have a safety phone call 12 weeks between in-person clinic visits until 90 days after commercial drug is available post regulatory approval or until study termination.

The primary endpoint of the main study is to evaluate the safety and tolerability of long-term dosing of losmapimod tablets in subjects with FSHD1. Secondary endpoints include assessment of target engagement of losmapimod in blood and skeletal muscle and repeated dose pharmacokinetics in subjects with FSHD1 over long-term dosing.

The extension will continue investigation of efficacy with assessment of skeletal muscle by ultrasound as well as the safety, tolerability, pharmacokinetics (PK), and exploration of efficacy measures including whole body skeletal muscle MRI and selected clinical outcome assessments during long- term dosing with losmapimod tablets in adult subjects with FSHD1. Secondary endpoints include assessment of efficacy as evaluated by whole body skeletal muscle MRI parameters, safety and tolerability of long-term dosing, target engagement of losmapimod in blood and skeletal muscle and repeated dose pharmacokinetics in subjects with FSHD1 over long-term dosing.

ELIGIBILITY:
Inclusion Criteria:

* FSHD1 subjects age 18-65 years.
* Subject will sign and date an informed consent form (ICF).
* Confirmed diagnosis of FSHD1 with 1 to 9 repeats via assessment of the size of the D4Z4 array on chromosome 4. Genetic confirmation must be obtained prior to the screening MRI and baseline muscle biopsy; genetic confirmation can come from previous testing if verified with appropriate documentation.
* Must be willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, scheduled needle muscle biopsies, and other study procedures.
* Both male and female subjects must be willing to practice an approved method of birth control.
* Clinical Severity Score between 2 and 4 on Ricci's Scale (scale range is from 0 to 5). Subjects that use a wheelchair or walker for any activity are not permitted to enroll in the study.
* Commitment to complete the 2 visits for skeletal muscle needle biopsy and all visits for whole-body MRI.
* Able to complete the RWS, TUG, and FSHD PROs (FSHD-RODS and FSHD-HI) at the screening visit.
* Must have an MRI-eligible muscle for biopsy as determined by the central reader.
* Subject must complete the main study through the Week 60 visit in order to participate in the open-label extension study.

Exclusion Criteria:

* History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include, but is not limited to, history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; history or presence of clinically significant pathology; clinically significant history of mental disease; and history of cancer, except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ (all 3 with no recurrence for the last 5 years).
* Subject has a known or clinically suspected infection with human immunodeficiency virus or hepatitis B or C viruses.
* Subject has current clinically significant liver (alanine aminotransferase > 2X upper limit of normal or total bilirubin >1.5 X upper limit of normal) or kidney (GFR < 30 mL/min/1.73m2) dysfunction.
* Subject screens positive for hepatitis B surface antigen, hepatitis C virus (HCV) antibody, or antibodies against human immunodeficiency viruses 1 and 2 (HIV 1/HIV 2 antibodies).
* Subject has any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, or other gastrointestinal tract surgery, except appendectomy).
* Subject has a standard 12-lead ECG demonstrating QT interval by Fredericia (QTcF) >450 msec for male subjects and QTcF >470 msec for female subjects at Screening. If QTcF exceeds 450 msec for males or 470 msec for females, the ECG will be repeated 2 more times, and the average of the 3 QTcF values will be used to determine the subject's eligibility.
* Subject has a history of cardiac dysrhythmias requiring anti-arrhythmia treatment(s); or history or evidence of abnormal ECGs that, in the opinion of the investigator or Medical Monitor, would preclude the subject's participation in the study.
* Male subject has a female partner who is planning to become pregnant during the study or within 90 days after the last study drug dose.
* Subject has donated blood (of approximately 1 pint [500 mL] or more) or has had any significant loss of blood within 90 days before the first study drug dose, as determined by the investigator.
* Vaccination with a live attenuated vaccine within 6 weeks of randomisation.
* Subject has a history of alcohol, analgesic/opioid, and/or illicit drug abuse as defined by the American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, in the last 6 months before screening, or a positive test for drugs of abuse at screening.
* Subject has participated in a clinical trial in which they have received an investigational product within the following time period prior to enrolment in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever was longer).
* For subjects that are on drug(s) or supplements that may affect muscle function as determined by the treating physician or included in the list of drugs presented in Section 15: subjects must be on a stable dose of that drug(s) or supplement for at least 3 months prior to enrollment in the study and remain on that stable dose for the duration of the study (list of drugs presented in Section 15). Changes to the dose or treatment discontinuation during the study can only be done for strict medical reasons by the treating physician with clear documentation and notification to the Sponsor.
* Subject has a history of sensitivity to any of the study medications or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicated their participation.
* Female subject is pregnant as determined by positive urine Human Chorionic Gonadotropin (HCG) test at Screening or prior to dosing.
* Female subject is lactating.
* Subject is unwilling or unable to follow the procedures outlined in the protocol.
* Subject has any contraindication for MRI (including severe claustrophobia and any shrapnel or metal implants in the body that are not MRI compatible).
* Subject was mentally or legally incapacitated up to 2 years prior to enrollment.
* Subject has abnormal laboratory results indicative of any significant medical disease that, in the opinion of the investigator or the medical monitor, would preclude the subject's participation in the study.
* Subject, or close relative of the subject, is the investigator or a subinvestigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study at that site.
* Subject has taken any anticoagulants for at least 1 month and anti-platelet agents for at least 1 week before each muscle biopsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour AM, Sarov-Blat L, Cai G, Fossler MJ, Sprecher DL, Graggaber J, McGeoch AT, Maison J, Cheriyan J. Safety, tolerability, pharmacokinetics and pharmacodynamics of losmapimod following a single intravenous or oral dose in healthy volunteers. Br J Clin Pharmacol. 2013 Jul;76(1):99-106. doi: 10.1111/bcp.12063. PMID 23215699
- [Background] Cheriyan J, Webb AJ, Sarov-Blat L, Elkhawad M, Wallace SM, Maki-Petaja KM, Collier DJ, Morgan J, Fang Z, Willette RN, Lepore JJ, Cockcroft JR, Sprecher DL, Wilkinson IB. Inhibition of p38 mitogen-activated protein kinase improves nitric oxide-mediated vasodilatation and reduces inflammation in hypercholesterolemia. Circulation. 2011 Feb 8;123(5):515-23. doi: 10.1161/CIRCULATIONAHA.110.971986. Epub 2011 Jan 24. PMID 21262998
- [Background] de Greef JC, Frants RR, van der Maarel SM. Epigenetic mechanisms of facioscapulohumeral muscular dystrophy. Mutat Res. 2008 Dec 1;647(1-2):94-102. doi: 10.1016/j.mrfmmm.2008.07.011. Epub 2008 Aug 3. PMID 18723032
- [Background] Han JJ, Kurillo G, Abresch RT, de Bie E, Nicorici A, Bajcsy R. Reachable workspace in facioscapulohumeral muscular dystrophy (FSHD) by Kinect. Muscle Nerve. 2015 Feb;51(2):168-75. doi: 10.1002/mus.24287. Epub 2014 Nov 19. PMID 24828906
- [Background] Statland JM, Tawil R. Risk of functional impairment in Facioscapulohumeral muscular dystrophy. Muscle Nerve. 2014 Apr;49(4):520-7. doi: 10.1002/mus.23949. Epub 2014 Feb 10. PMID 23873337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center, open-label pilot study that investigated the safety, tolerability, pharmacokinetic (PK), and target engagement during long-term dosing with losmapimod tablets in adult participants with facioscapulohumeral muscular dystrophy 1 (FSHD1). The study comprised of a main study and an extension phase. A total of 14 participants were enrolled.
Pre-assignment Details: Participants were administered 15 milligrams (mg) losmapimod orally twice-daily (BID) for approximately 1 year during the main study and had the option to roll over into the extension study and continued to receive the treatment. The Sponsor decided to terminate the extension phase because the primary endpoint of Phase 3 REACH (NCT05397470) was not achieved.
Groups:
- Losmapimod 15 Milligrams (mg) Twice Daily (BID): Participants were administered Losmapimod 15 mg twice-daily (BID) orally for approximately one year and then rolled over to extension phase to receive Losmapimod at the same dose until 90 days after commercial drug is available post regulatory approval or study termination.
Period: Main Study Phase (Up to 52 Weeks)
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Started | 14
Completed | 14
Not Completed | 0
Period: Extension Phase (Up to 68 Weeks)
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Started | 12
Completed | 0
Not Completed | 12
Not completed — Sponsor terminated OLE as REACH (NCT05397470) Phase 3 study in FSHD did not meet primary endpoint. | 12

BASELINE CHARACTERISTICS:
Population: Safety analysis set which comprised of participants who received at least one dose of losmapimod.
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A TEAE is an AE that begins on or after the first dose of study drug and before the stop of study drug + 7 days or begins before the first dose of study drug and worsens on or after the first dose of study drug and before the stop of study drug + 7 days. A Serious adverse event (SAE) is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to 68 Weeks
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 14
Participants
  Any TEAE | 14
  Any serious TEAE | 2

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Chemistry Parameters
Description: Blood samples were collected for the analysis of chemistry parameters: Glucose, sodium, potassium, calcium, inorganic phosphate, total protein, albumin, blood urea nitrogen, creatinine, uric acid, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, lactate dehydrogenase and creatine phosphokinase.
Time Frame: Up to 68 Weeks
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 14
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters: hemoglobin (including mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration), hematocrit, red blood cell count, total white blood cell count, platelet count. Differential blood counts, including basophils, eosinophils, neutrophils, lymphocytes, and monocytes
Time Frame: Up to 68 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 14
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Serum Coagulation Parameters
Description: Blood samples were collected for the analysis of Serum coagulation parameters: International normalized ratio, prothrombin time, activated partial thromboplastin time and fibrinogen.
Time Frame: Up to 68 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 14
Participants | 0

5. Secondary Outcome: Percent Change From Baseline in the Ratio of Phosphorylated HSP27 (pHSP27) /Total HSP27 in Sorbitol-stimulated Whole Blood
Description: Phosphorylated HSP27 in peripheral whole blood with ex-vivo sorbitol stimulation and in skeletal muscle (without sorbitol stimulation) was measured at specified time points. The pre-treatment value was considered as Baseline for change from Baseline calculations. The geometric mean for fold percent change from Baseline (and 95% confidence interval) in pHSP27/total HSP27 was calculated. Percent change from baseline = 100*(exp(mean of change from baseline on the log-transformed scale) - 1).
Time Frame: Baseline and at Week 44
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 11
Percent change | -48.3 [-55.4 to -40.1]

6. Secondary Outcome: Percent Change From Baseline in Ratio of pHSP27/Total HSP27 in Muscle
Description: Phosphorylated HSP27 in skeletal muscle (without sorbitol stimulation) was measured at specified time points. The pre-treatment value was considered as Baseline for change from Baseline calculations. The geometric mean for fold percent change from Baseline (and 95% confidence interval) in pHSP27/total HSP27 was calculated. Percent change from baseline = 100*(exp(mean of change from baseline on the log-transformed scale) - 1).
Time Frame: Baseline and at Week 8
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 2
Percent change | 33.9 [-78.3 to 726.5]

7. Secondary Outcome: Plasma Concentration of Losmapimod
Description: Blood samples were collected to measure the plasma concentration of losmapimod at specified timepoints.
Time Frame: Post-dose at Baseline, Week 4, Week 8, Week 20, Week 32, Week 44, and Week 56
Population: Safety Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 12
Nanograms per milliliter
  Baseline | 58.923 (0.488)
  Week 4: number analyzed (Participants) | 6
  Week 4 | 92.737 (0.220)
  Week 8: number analyzed (Participants) | 2
  Week 8 | 83.006 (0.356)
  Week 20: number analyzed (Participants) | 7
  Week 20 | 80.889 (0.315)
  Week 32: number analyzed (Participants) | 7
  Week 32 | 82.261 (0.275)
  Week 44 | 75.029 (0.316)
  Week 56 | 66.268 (0.367)

8. Secondary Outcome: Muscle Concentration of Losmapimod
Description: Muscle biopsies were collected to measure the concentration of losmapimod at specified timepoints.
Time Frame: Post dose at Baseline, Week 4, Week 8 and Week 44
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 6
Nanograms per milliliter
  Baseline: number analyzed (Participants) | 5
  Baseline | 0.215 (0.348)
  Week 4 | 84.456 (0.198)
  Week 8: number analyzed (Participants) | 2
  Week 8 | 77.904 (0.134)
  Week 44: number analyzed (Participants) | 3
  Week 44 | 73.193 (0.199)

ADVERSE EVENTS:
Time Frame: Up to 68 Weeks
Description: TEAEs and serious TEAEs were collected in Safety population which included all participants who received study drug.
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 15 Milligrams (mg) Twice Daily (BID) (N=14)
Pneumonia (Infections and infestations) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 15 Milligrams (mg) Twice Daily (BID) (N=14)
Palpitations (Cardiac disorders) | 2
Middle ear effusion (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 3
Eczema eyelids (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Colitis microscopic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Feeling cold (General disorders) | 1
Influenza like illness (General disorders) | 3
Non-cardiac chest pain (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 10
Cystitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 7
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Onychomycosis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Oral infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Epicondylitis (Injury, poisoning and procedural complications) | 3
Face injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 8
Foreign body (Injury, poisoning and procedural complications) | 1
Heat stroke (Injury, poisoning and procedural complications) | 1
Inflammation of wound (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 2
Nerve injury (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Blood pressure diastolic increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 3
Neuralgia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Penile rash (Reproductive system and breast disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 6
Eczema (Skin and subcutaneous tissue disorders) | 6
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT04004000/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04004000/SAP_001.pdf